CLINICAL TRIAL: NCT04956601
Title: A Multicenter, Randomized, Controlled Trial of Adjuvant Radiotherapy in Patients With Early Endometrial Cancer Based on Moderate Risk Molecules Classification
Brief Title: Adjuvant Radiotherapy in Patients With Early Endometrial Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Junjie Wang, Peking University Third Hospital, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECART001
Record Dates: First submitted 2021-07-02; First posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Endometrial Cancer; Pathology; Radiotherapy
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VBT (Experimental): CT image guided high-dose-rate vaginal brachytherapy, 30Gy/6f, 2f/w.
  Interventions: Radiation: vaginal brachytherapy/pelvic external beam radiotherapy
- EBRT (Active Comparator): Pelvic external beam radiotherapy，IMRT/VAMT，IGRT suggested，DT 45Gy/25f.
  Interventions: Radiation: vaginal brachytherapy/pelvic external beam radiotherapy

INTERVENTIONS:
Radiation: vaginal brachytherapy/pelvic external beam radiotherapy — high-dose-rate vaginal brachytherapy; pelvic external beam radiotherapy
  Other Names: Pelvic external beam radiotherapy

SUMMARY:
To compare the effect of vaginal brachytherapy as adjuvant treatment after operation when compared to pelvic external beam radiotherapy in patients with early endometrial cancer based on moderate risk molecules classification.

DETAILED DESCRIPTION:
After being informed the study and potential risk，all patients giving written informed consent will be undergo a 1-week screening period determine eligibility for study entry. At week 0, patients who meet the eligibility will be randomized in a 1:1 ratio to vaginal brachytherapy or pelvic external beam radiotherapy. After treatment, patients were followed up regularly.

ELIGIBILITY:
Inclusion Criteria:

1. Endometrial adenocarcinoma is confirmed by pathology, and the molecular types were microsatellite instability type and low copy type;
2. Stage IA and grade 3 or stage IB (FIGO 2009), without substantial lymph-vascular space invasion;
3. Surgery must have included a hysterectomy and bilateral adnexectomy. Pelvic lymph node sampling and para-aortic lymph node sampling are optional;
4. ECOG score is 0-2;
5. The interval time between surgery and radiotherapy is no more than 8 weeks;
6. The routine blood examination was normal;
7. Compliance is good and informed consent is voluntarily signed.

Exclusion Criteria:

1. The patients receive chemotherapy;
2. History of previous malignant disease;
3. Previous diagnosis of Crohn's disease or ulcerative colitis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
DFS | 5-year
  disease-free survival from being received treatment

SECONDARY OUTCOMES:
Failure mode | 5-year
  vaginal recurrences; pelvic recurrence; distant metastases
OS | 5-year
  Overall survival from being received treatment
Toxicities | 5-year
  from being received treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University 3rd Hospital, Beijing, Beijng, China

IPD SHARING:
Plan to Share IPD: Undecided